CLINICAL TRIAL: NCT07112430
Title: Intranasal Fentanyl to Reduce Pain Intensity Associated With Retinopathy of Prematurity Screening in Preterm Infants: A Randomized Control Trial
Brief Title: Fentanyl Intranasal for Retinopathy of Prematurity Screening in Preterm Infants
Acronym: FIREFLY
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: IWK Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IWK_INF_PainTrial2025
Record Dates: First submitted 2025-07-29; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-06

CONDITIONS: Neonatal Pain; Retinopathy of Prematurity (ROP); Pain Management; Infant, Premature; Fentanyl; Infant, Newborn; Neonatal Intensive Care Units; Analgesia; Intranasal Drug Administration
Keywords: intranasal fentanyl; fentanyl; neonatal analgesia; procedural pain; ROP screening; Retinopathy of Prematurity; Preterm infants; Premature infants; infant pain; Non-invasive analgesia; Opioid analgesia; Intranasal drug delivery; Neonatal intensive care; NICU; Pain management in neonates; Infant procedural sedation
MeSH Terms: conditions — Retinopathy of Prematurity; Agnosia; Premature Birth; Pain, Procedural | interventions — Fentanyl; Saline Solution

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled, parallel-group trial. Eligible preterm infants undergoing their first retinopathy of prematurity (ROP) screening will be randomly assigned to receive either intranasal fentanyl or a placebo (normal saline) prior to the procedure. Each participant will remain in their assigned group for the duration of the intervention. The primary aim is to evaluate the analgesic effectiveness and safety of intranasal fentanyl compared to placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a quadruple-masked (participant, care provider, investigator, and outcome assessor) randomized controlled trial. Blinding is maintained through the use of identical-appearing administration devices for the study drug and placebo. The clinical team, including those administering the intervention and assessing outcomes such as PIPP-R scores, are unaware of group allocation to reduce bias. Allocation concealment is ensured via centralized randomization and pharmacy-controlled preparation of interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intranasal Fentanyl Group (Experimental): Participants in this group will receive intranasal fentanyl at a dose of 2 mcg/kg administered 5 minutes prior to initiation of retinopathy of prematurity (ROP) screening. Fentanyl will be delivered via a mucosal atomization device in conjunction with standard non-pharmacologic comfort measures.
  Interventions: Drug: Fentanyl Citrate (Intranasal)
- Placebo Group (Placebo Comparator): Participants in this group will receive an equivalent volume of intranasal normal saline (placebo) administered 5 minutes prior to ROP screening using a mucosal atomization device. Standard non-pharmacologic comfort measures will also be provided.
  Interventions: Drug: Normal Saline (Placebo, Intranasal)

INTERVENTIONS:
Drug: Fentanyl Citrate (Intranasal) — Fentanyl citrate will be administered intranasally at a dose of 2 mcg/kg via a mucosal atomization device, 5 minutes prior to ROP screening. Used in conjunction with standard non-pharmacologic comfort strategies.
  Arms: Intranasal Fentanyl Group
Drug: Normal Saline (Placebo, Intranasal) — An equivalent volume of intranasal normal saline will be administered using a mucosal atomization device, 5 minutes prior to ROP screening.
  Arms: Placebo Group

SUMMARY:
This single-center, double-blinded, randomized controlled trial aims to evaluate the efficacy and safety of intranasal fentanyl (INF) for reducing pain during retinopathy of prematurity (ROP) screening in preterm infants. The trial will enroll preterm neonates (≤32 weeks gestation) requiring ROP screening and randomize them to receive either intranasal fentanyl (2 mcg/kg) or a placebo (normal saline) 5-10 minutes prior to the procedure. The primary outcome is pain intensity measured using the Premature Infant Pain Profile-Revised (PIPP-R) at 30 seconds after speculum insertion. Secondary outcomes include physiological (heart rate, oxygen saturation), behavioral (crying time), and recovery indicators, along with adverse events and need for rescue dosing. This study addresses a critical gap in evidence by exploring a non-invasive pharmacologic intervention for procedural pain in the neonatal intensive care unit (NICU) setting. The findings may inform future practice and guidelines for neonatal pain management.

DETAILED DESCRIPTION:
This double-blinded, randomized controlled trial will evaluate the effectiveness and safety of intranasal fentanyl (INF) in reducing procedural pain associated with retinopathy of prematurity (ROP) screening in preterm infants. ROP screening is a necessary but painful procedure routinely performed in neonatal intensive care units (NICUs), and there remains a lack of consistent and effective pharmacological strategies for managing associated pain, particularly in preterm infants.

Eligible participants will include preterm infants born at or before 32 weeks gestation and scheduled for their first ROP exam. Infants with congenital anomalies, hemodynamic instability, or contraindications to fentanyl will be excluded. Participants will be randomized in a 1:1 ratio to receive either intranasal fentanyl (2 mcg/kg) or an equivalent volume of intranasal saline placebo. Randomization will be stratified by gestational age (<28 weeks vs. ≥28 weeks) to ensure balance between treatment arms.

The intervention will be administered 5-10 minutes prior to the ROP screening using a mucosal atomization device to optimize nasal absorption and bioavailability. Non-pharmacological comfort measures such as swaddling and non-nutritive sucking will be applied uniformly to all participants as standard of care. The ROP examination will be performed by a pediatric ophthalmologist using a standardized protocol including use of a speculum and scleral depression.

The primary outcome is pain intensity as measured by the Premature Infant Pain Profile-Revised (PIPP-R) at 30 seconds after speculum insertion. Secondary outcomes include additional PIPP-R scores at subsequent timepoints (e.g., speculum removal), changes in physiological parameters (heart rate, oxygen saturation), crying time, pain recovery trajectory, and the occurrence of any adverse events such as respiratory depression, apnea, or need for rescue dosing.

Vital signs and continuous cardiorespiratory monitoring will be conducted before, during, and after the procedure to identify any immediate adverse effects. Pain scoring will be conducted by trained, blinded assessors who are not involved in administering the intervention or performing the ROP exam.

Safety monitoring will include predefined criteria for adverse events and a data safety monitoring plan, including interim review by an independent neonatologist. Any infant experiencing a serious adverse event will be promptly evaluated, and unblinding may occur if necessary for clinical care.

This trial is designed to address a significant gap in neonatal pain management by generating high-quality evidence on the feasibility, safety, and efficacy of intranasal fentanyl in a vulnerable population. The use of a non-invasive, easily administered opioid analgesic could improve procedural pain control without introducing the risks associated with intravenous access. Findings from this study may inform neonatal pain management protocols and support the development of evidence-based guidelines for the use of intranasal fentanyl in NICU settings.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at <32 weeks gestational age
* Undergoing their first screening for retinopathy of prematurity (ROP)
* Clinically stable at the time of the procedure
* Parental or legal guardian informed consent obtained

Exclusion Criteria:

* Known or suspected congenital anomalies affecting the nose
* Receipt of systemic analgesics or sedatives at the time of ROP screening
* Nasal obstruction or malformations that interfere with intranasal drug delivery
* Contraindications to fentanyl (e.g., known hypersensitivity)

Ages: 30 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity during ROP screening | 30 seconds after speculum insertion during ROP screening
  Pain intensity will be measured using the Premature Infant Pain Profile-Revised (PIPP-R) score. The score will be assessed 30 seconds after insertion of the speculum, during the ROP eye examination.

SECONDARY OUTCOMES:
Proportion of infants with low to mild pain | 30 seconds after speculum insertion
  The proportion of infants experiencing low or mild pain will be assessed using the PIPP-R score, with established thresholds to categorize pain levels. Scores will be assigned by blinded assessors reviewing synchronized video recordings.
Pain response during ROP screening | Every 30 seconds throughout the procedure
  Pain scores will be measured using PIPP-R at 30-second intervals from speculum insertion until the end of the ROP screening to evaluate procedural pain trajectory. Scores will be coded from video by blinded assessors.
Pain recovery following ROP screening | End of procedure, 1-minute and 5-minutes post-procedure
  PIPP-R scores will be used to evaluate pain recovery immediately at procedure end, and at 1- and 5-minutes post-procedure. This will assess the time course of pain resolution.
Cry time during and after procedure | During and after the ROP screening procedure
  Total cry time and first cry duration (in seconds) will be measured from video recordings of the procedure, assessed by trained, blinded coders.
Salivary cortisol levels | Pre-procedure and 20 minutes post-procedure
  Salivary cortisol (μg/dL), a hormonal marker of stress, will be measured before the procedure and 20 minutes after to assess endocrine pain response.
Adverse events related to intervention | During procedure and up to 4 hours post-intervention
  Safety will be evaluated by monitoring predefined adverse events such as apnea, bradycardia, hypotension, chest rigidity, desaturation, feeding intolerance, need for airway support, and inadequate pupil dilation.
Duration of ROP examination | Entire ROP procedure from speculum insertion to removal
  Total duration of the ROP exam will be recorded in seconds from speculum insertion to removal using timestamped video to assess procedural efficiency.
Physiological pain indicators (Heart rate) | Baseline, 30 seconds after speculum insertion, 1-minute and 5-minutes post-procedure
  Changes in heart rate (beats per minute) will be measured as physiological correlates of pain. Data will be collected before, during, and after the procedure.
Physiological pain indicators (RR) | Baseline, 30 seconds after speculum insertion, 1-minute and 5-minutes post-procedure
  Changes in respiratory rate (breaths per minute) will be measured as physiological correlates of pain. Data will be collected before, during, and after the procedure.
Physiological pain indicators (blood pressure) | Baseline, 30 seconds after speculum insertion, 1-minute and 5-minutes post-procedure
  Changes in blood pressure (mmHg) will be measured as physiological correlates of pain. Data will be collected before, during, and after the procedure.
Physiological pain indicators (Oxygen saturation) | Baseline, 30 seconds after speculum insertion, 1-minute and 5-minutes post-procedure
  Changes in oxygen saturation (SpO₂) will be measured as physiological correlates of pain. Data will be collected before, during, and after the procedure.

IPD SHARING:
Plan to Share IPD: Undecided
The plan to share individual participant data (IPD) is currently undecided. IPD sharing may be considered in the future depending on institutional policies, ethics approval, and participant consent. If data sharing is pursued, it will involve de-identified data underlying published results, and appropriate data use agreements and secure access mechanisms will be established. No final decision has been made at this stage.